CLINICAL TRIAL: NCT01976182
Title: Prospective, Sequential Multiple Assignment, Multicentric, Phase II Randomized Controlled Trial on Two Parallel Groups Comparing the Efficacy of Two Immunosuppressive Drugs (methotrexate, Cyclophosphamide) in Large Granular Lymphocytes Leukemia
Brief Title: Prospective, Multicentric, Phase II Randomized Controlled Trial on Two Parallel Groups Comparing the Efficacy of Two Immunosuppressive Drugs (methotrexate, Cyclophosphamide) in Large Granular Lymphocytes Leukemia
Acronym: LGL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC12_8972 _LGL
Record Dates: First submitted 2013-10-22; First posted 2013-11-05 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Large Granular Lymphocytes Leukemia
Keywords: large granular lymphocytes leukemia; immunosuppressive drugs; methotrexate; cyclophosphamide; efficiency; phase II randomized controlled trial
MeSH Terms: interventions — Methotrexate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- METHOTREXATE (Active Comparator): In step 1, 55 patients will receive methotrexate 10mg / m² orally once a week, (at split doses of 5 mg/m2 in the morning and 5 mg/m2 at night), that is to say 2 tablets of 2.5 mg at each take
  In step 2, responders at Month 4 (CR or PR) will be treated during 8 additional months with methotrexate at the same dosage.
  Non responders at Month 4 will be randomized and treated either by:
  * Cyclophosphamide delivered at 100 mg orally once daily, that is to say 2 tablets of 50 mg at each take between Month 5 and Month 8, decreased to 50 mg orally once daily beyond Month 8 for responders at Month 8;
  * Ciclosporine A delivered at 3 mg/kg per day (at split doses of 1.5 mg/kg in the morning and 1.5 mg/kg at night) orally administered.
  Interventions: Drug: Methotrexate
- CYCLOPHOSPHAMIDE (Active Comparator): In step 1, 55 patients will receive cyclophosphamide 100 mg orally once daily, that is to say 2 tablets of 50 mg at each take.
  In step 2, responders at Month 4 (CR or PR) will be treated during 8 additional months with cyclophosphamide (at 50 mg orally once daily);
  Non responders at Month 4 will be randomized and treated either by:
  * Methotrexate administered at 10 mg/m2 orally once a week (at split doses of 5 mg/m2 in the morning and 5 mg/m2 at night), that is to say 2 tablets of 2.5 mg at each take;
  * Ciclosporine A delivered at 3 mg/kg per day (at split doses of 1.5 mg/kg in the morning and 1.5 mg/kg at night) orally administered.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Methotrexate — methotrexate 10mg / m² orally once a week, (at split doses of 5 mg/m2 in the morning and 5 mg/m2 at night), that is to say 2 tablets of 2.5 mg at each take, during 4 months.
  Arms: METHOTREXATE
Drug: Cyclophosphamide — cyclophosphamide 100 mg orally once daily, that is to say 2 tablets of 50 mg at each take, during 4 months.
  Arms: CYCLOPHOSPHAMIDE

SUMMARY:
LGL leukemia represents a rare subtype of chronic T or NK lymphoproliferative disorders. It is an indolent disease, the main hematological or autoimmune complications lead to a treatment in more than 60% of patients.

Investigators set up at the University Hospital of Rennes, a database of more than 300 patients with LGL leukemia from major French services that support this disease, and published in 2010 the largest series of patients in the world (n = 229). However, the limited heterogeneity and retrospective data collected, as all previously released, makes it difficult the proposal of consensual treatment options. If first and second line treatments are based on the use of immunosuppression with methotrexate, cyclophosphamide, or cyclosporin A, no molecule has proven superiority over others. Methotrexate and cyclophosphamide are mainly used in the first line. Invetigators just have in the literature data on about 100 patients treated with either of these drugs. Combining the results of our series with those in the literature, invetigators estimate the respective overall response rate (RG) and complete response rate (CR) in 55% and 30% for methotrexate, and 60% and 50% for cyclophosphamide.

Thus, there are four objective in this study :

1. to compare the respective efficacies of methotrexate and cyclophosphamide when administered as first-line therapies in patients suffering from T/NK LGL leukemia with severe neutropenia or neutropenia associated with infections, and/or anemia requiring transfusions, and/or auto-immune associated disease
2. to evaluate the percentage of patients refractory to methotrexate or cyclophosphamide for which a second line treatment is efficacious
3. to explore, in case of non-response to the first-line therapy, the efficacy of ciclosporine A, the comparison being performed with the treatment which was not administered in the first-line therapy
4. to evaluate the response rate according to the phenotypic subtype of LGL leukemia.

DETAILED DESCRIPTION:
Large Granular Lymphocyte (LGL) leukemia is a clonal disorder involving tissue invasion of marrow, spleen and liver. Clinical presentation is dominated by recurrent infections associated with neutropenia, anemia, splenomegaly, and auto-immune diseases, particularly rheumatoid arthritis. Both T cell and NK cell subtypes of LGL leukemia are indolent disease and considered as a chronic illness and lead to a treatment in more than 60% of patients.

LGL leukemia displays a chronic clinical course. Recommendations regarding therapy are similar for both subtypes. Indications for treatment include 1) severe neutropenia (ANC <500 mm3); 2) neutropenia (ANC <1500mm3) with symptomatic recurrent infections; 3) symptomatic or transfusion-dependent anemia and 4) associated autoimmune conditions requiring therapy, most often rheumatoid arthritis.

There is no standard treatment for patients with LGL leukemia. The numerous case reports published do not provide a consensus for a particular treatment. All the six largest series published in the literature so far (collecting data on more than 40 patients) are retrospective.

Immunosuppressive therapy remains the foundation of treatment including single three agents i.e. methotrexate, oral cyclophosphamide and ciclosporin A. However prospective trials involving large numbers of patients have not been performed and no molecule has proven superiority over others.

Invetigators set up at the University Hospital of Rennes, a database of more than 300 patients with LGL leukemia from major French services that support this disease, and published in 2010 the largest series of patients in the world (n = 229). However, the limited heterogeneity and retrospective data collected, as all previously released, makes it difficult the proposal of consensual treatment options. Combining the results of our series with those of the literature, invetigators estimate that overall response rate and complete response rate are 55% and 30% with methotrexate, 60% and 50% with cyclophosphamide, and 55% and less than 20% with ciclosporine A, respectively.

Thus, there are four objective in this study :

1. to compare the respective efficacies of methotrexate and cyclophosphamide when administered as first-line therapies in patients suffering from T/NK LGL leukemia with severe neutropenia or neutropenia associated with infections, and/or anemia requiring transfusions, and/or auto-immune associated disease
2. to evaluate the percentage of patients refractory to methotrexate or cyclophosphamide for which a second line treatment is efficacious
3. to explore, in case of non-response to the first-line therapy, the efficacy of ciclosporine A, the comparison being performed with the treatment which was not administered in the first-line therapy
4. to evaluate the response rate according to the phenotypic subtype of LGL leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Common criteria of LGL leukemia: the diagnosis is based on a chronic LGL peripheral blood expansion (>0.5x109/L), usually lasting more than 6 months
* Specific criteria for T-LGL leukemia or NK-LGL lymphocytosis or chronic NK-LGL leukemia:

  * Specific criteria for T-LGL leukemia:
* Expression of LGL surface markers compatible with an activated T-cell (commonly alpha-beta+/CD3+/CD8+/CD57+ and/or CD16+) phenotype or gamma-delta+ T cells;
* Clonal rearrangement of TCRγ gene using PCR or specific and clonal Vβ expression using FCM.

  * Specific criteria for NK-LGL lymphocytosis or chronic NK LGL leukemia:
* Expression of LGL surface markers compatible with a NK cell (commonly CD3-/CD8+/CD16+ and/or CD16+/CD56+) phenotype;
* CD56+ or CD16+ NK cells greater than 0.75x109/L;
* The term of chronic NK-LGL lymphocytosis is used for patients with chronic illness (NB: patients with massive tissue LGL infiltration of the spleen, liver and bone marrow and presenting aggressive clinical behavior are considered as having aggressive NK-LGL leukemia and should not be included).
* Age above 18 years
* ECOG performance status of 0-2
* Life expectancy of at least 1 year
* Lack of previous treatment (except with G-CSF or transfusions)
* At least one indication of treatment:

  * Isolated severe neutropenia (ANC <0.5x109/L) or neutropenia (ANC <1.5x109/L) with two or more infections requiring antibiotics;
  * Anemia (whatever the underlying mechanism: pure red cell aplasia or marrow infiltration) requiring transfusions greater than 2 units for two months prior to inclusion, or symptomatic anemia (hemoglobin <10g/dl) with impairment of the quality of life;
  * Associated complications such as systemic diseases or auto-immune diseases (i.e. recurrent uveitis, cutaneous vasculitis, autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura, rheumatoid arthritis resistant to steroids and/or immunomodulator agents (colchicin, disulone, hydrochloroquine)) and justifying a treatment with methotrexate or cyclophosphamide
* Written informed consent

Exclusion Criteria:

* Inability to understand or to follow study procedures
* Prior or concurrent malignancy within the past 5 years except inactive nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Other serious medical illnesses, such as hepatic, renal, cardiac, pulmonary, neurologic, or metabolic disease that would preclude the patient's ability to tolerate methotrexate, cyclophosphamide, or ciclosporine A
* Reactive LGL lymphocytosis (i.e. after viral infection)
* ALAT/ASAT or alkalin phosphatases >3 times normal values
* Creatinine clairance <50 ml/min
* Serologic evidence of HIV, hepatitis C or hepatitis B infection
* Non effective contraception
* Positive pregnancy test
* Nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) | at Month 4
  The main endpoint will be the hematological CR rate evaluated after 4 months of treatment (binary endpoint). Complete response (CR) is defined as a normalization of clinical examination (disappearance of splenomegaly) and a complete normalization of blood counts (i.e., hemoglobin >12g/dL, platelets >150x109/L, ANC >1.5x109/L), lymphocytosis <4x109/L and circulating LGL in the normal range (<0.3x109/L). The number of LGL will be quantitated on blood smears.

SECONDARY OUTCOMES:
overall response rate (ORR) | at Month 4, and at Month 8 and Month 12 in non-responders at Month 4
  Hematological overall response rate (ORR) defined as the sum of complete responses and partial responses over the total number of patients.
Complete response (CR) | at Month 8 and Month 12
  Complete response (CR) is defined as a normalization of clinical examination (disappearance of splenomegaly) and a complete normalization of blood counts (i.e., hemoglobin >12g/dL, platelets >150x109/L, ANC >1.5x109/L), lymphocytosis <4x109/L and circulating LGL in the normal range (<0.3x109/L). The number of LGL will be quantitated on blood smears.
Hematological partial response (PR) | at Month 4, Month 8 and Month 12
  Hematological partial response (PR) defined as an improvement in blood counts which do not meet criteria for complete remission (e.g., ANC increasing more than 50% and reaching more than 0.5 but less than 1.5x109/L with non-recurrence of infections, or hemoglobin level increasing more than 2 g/dL from baseline and transfusion requirements stopping without normalization of the hemoglobin level defined as hemoglobin >12g/dL).
Progressive disease | at Month 4, Month 8 and Month 12
  Progressive disease defined as worsening of cytopenia or organomegaly or incidence of infections.
Time-to-relapse | from Month 4 to endpoint (in first-line treatment responders)
  Time-to-relapse (censored variable). Relapse is defined as re-occurrence of either neutropenia or anemia (ANC <1x109/L and/or hemoglobin <10g/dL) or clonal LGL >0.5x109/L in complete responders, or as a return to baseline values of either ANC or hemoglobin in partial responders, at two monthly consecutive blood tests.
Time-to-relapse | from Month 8 to endpoint (in second-line treatment responders)
  Time-to-relapse (censored variable). Relapse is defined as re-occurrence of either neutropenia or anemia (ANC <1x109/L and/or hemoglobin <10g/dL) or clonal LGL >0.5x109/L in complete responders, or as a return to baseline values of either ANC or hemoglobin in partial responders, at two monthly consecutive blood tests.
Molecular remission | at Month 4 and Month 12 for hematological complete responders
  Molecular remission defined as the disappearance of the clonal pattern of TCR gamma multiplex rearrangement and Phenotypic remission is defined as :
  * For the T subtype: disappearance of the excess of CD3+/CD8+ cells (or disappearance of the LGL clone according to the specific subtype observed at inclusion);
  * For the NK subtype: disappearance of the excess of CD3-/CD56+ cells (or disappearance of the LGL clone according to the specific subtype observed at inclusion)
Adverse events rate | Month 2, Month 4, Month 6, Month 8, Month 10, Month 12
  Adverse events rate
Compliance | Month 2, Month 4, Month 6, Month 8, Month 10, Month 12
  Compliance
relationship between the response to treatment and the phenotypic subtype | Day 1
  Identification of a relationship between the response to treatment and the phenotypic subtype characterized by the panel of monoclonal antibodies defined in the ancillary study subsection.

CONTACTS AND LOCATIONS:
Locations (59):
- France (59):
  - CHU Sud, Amiens
  - CHU Angers, Angers
  - Intern medecine Service - CH Antibes-Juan-les-Pins, Antibes
  - Hematology Service - CH Avignon, Avignon
  - Hematology Service - CH de la cote basque, Bayonne
  - hematology service - CH Beauvais, Beauvais
  - Hematology Service - CH Jean Minjoz, Besançon
  - Hematology Service - CH Beziers, Béziers
  - Hematology Unit - HOpital Avicienne, Bobigny
  - Hematology Service - CH Docteur Duchenne, Boulogne-sur-Mer
  - Hematology Service - CH de Brest, Brest
  - Institut d'Hématologie de Basse Normandie, Caen
  - Hematology Service - CH François Baclesse, Caen
  - hematology Service - CH Louis Pasteur, Chartres
  - Centre Hospitalier de Cholet, Cholet
  - Hopital Inter-Armées Percy, Clamart
  - hematology Service - CHU Estaing, Clermont-Ferrand
  - Hematology Service - Civils hospital, Colmar
  - Hematology Service CHSF, Corbeil-Essonnes
  - CHU Henri Mondor Lymphoid Hemopathy Unit, Créteil
  - Hematology Unit CH Michalon, Grenoble
  - Hematology Unit CHD Vendée, La Roche-sur-Yon
  - Hematology Unit CH LE MANS, Le Mans
  - CH Robert Boulin, Libourne
  - Hematology Unit CHRU Lille, Lille
  - Hematology Unit CHU Dupuytren, Limoges
  - CH de Bretagne Sud, Lorient
  - Hematology Unit CHU La Conception, Marseille
  - Hematology Unit - Institut Paoli-Calmettes, Marseille
  - Hematology Unit CH Meaux, Meaux
  - Hematology Unit CH Notre Dame Bon Secours, Metz
  - Hematogy Unit CHU ST ELOI, Montpellier
  - Hematology Unit CH E.MULLER, Mulhouse
  - Internal Medicine - CHU Hotel Dieu, Nantes
  - Oncology Unit CH Antoine Lacassagne, Nice
  - hematology Unit CHU Caremeau, Nîmes
  - Hematology Unit - CHR Orleans, Orléans
  - Hematology Service - Hopital La Pitié Salpetrière, Paris
  - Hematology Unit - Hopital Hotel Dieu, Paris
  - Hematology Unit - Hopital Saint Antoine, Paris
  - AP-HP Hôpital Necker - Enfants Malades, Paris
  - Hematology Unit - Hopital Saint Louis, Paris
  - Hematology Unit Hopital Saint Jean, Perpignan
  - Hematology Service- CH Haut Leveque, Pessac
  - Hematology Unit CH LYON SUD, Pierre-Bénite
  - Hematology Unit CHU La Miletrie, Poitiers
  - Hematology Unit CH René DUBOS, Pontoise
  - CH Annecy - Hematology Service, Pringy
  - Hematology Unit- Hopital Robert Debré, Reims
  - Hematology Service - CHU of Rennes, Rennes
  - Hematology Unit - CH Becquerel, Rouen
  - CH Yves Lefoll, Saint-Brieuc
  - Oncology Unit - Institut de cancérologie de la Loire, Saint-Priest-en-Jarez
  - CH Saint Quentin Oncohematology, Saint-Quentin
  - Hematology Unit CHU Toulouse, Toulouse
  - Hematology Unit CHU Bretonneau, Tours
  - Hematology Unit Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Intern Medecine Unit CHBA, Vannes
  - Hôpital André Mignot Centre Hospitalier de Versailles, Versailles

IPD SHARING:
Plan to Share IPD: No